CLINICAL TRIAL: NCT05549154
Title: A Study on Prevention Strategies for CKD-SHPT and Related Complications Based on General Vitamin D Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJTU1AF2022LSK-320
Record Dates: First submitted 2022-09-01; First posted 2022-09-22 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Disease 5D; Secondary Hyperparathyroidism Due to Renal Causes; Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose vitamin D group (Experimental): Vitamin D2 softgels 50,000 U/week
  Interventions: Drug: High-dose vitamin D2 softgels
- Low-dose vitamin D group (Experimental): low-dose vitamin D group
  Interventions: Drug: low-dose vitamin D2 softgels
- Control group (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: High-dose vitamin D2 softgels — 5000U/capsule of vitamin D2 soft capsule; High-dose VD group 50,000 U/week, 5 vitamin D2 softgels given twice a week each time; 25(OH)D > 80ng/ml after 3 months of intervention or within 3 months in both groups, changed to 5,000 U/ weekly maintenance until the full 6 months of intervention. To prevent unmasking, the maintenance dose was still given twice weekly (the first time 1 vitamin D2 capsule + 4 placebo capsules were given and the second time 5 placebo capsules were given)
  Arms: High-dose vitamin D group
Drug: low-dose vitamin D2 softgels — 5000U/capsule of vitamin D2 soft capsule; low-dose VD group 25,000 U/week, 3 vitamin D2 softgels + 2 placebo in the first dose, 2 vitamin D2 softgels + 3 placebo in the second dose, 25(OH)D > 80ng/ml after 3 months of intervention or within 3 months in both groups, changed to 5,000 U/ weekly maintenance until the full 6 months of intervention. To prevent unmasking, the maintenance dose was still given twice weekly (the first time 1 vitamin D2 capsule + 4 placebo capsules were given and the second time 5 placebo capsules were given);
  Arms: Low-dose vitamin D group
Drug: placebo — placebo was filled with excipients (aniseed ether, refined vegetable oil), and the shape and size were the same as vitamin D2 soft capsule.the control group was given placebo, 5 placebo capsules twice weekly for 6 months of the intervention. The medication was dispensed by a designated person (not the investigator) in advance and independently according to the patient's medication number (only the drug number was provided on the outer packaging).
  Arms: Control group

SUMMARY:
1. Study content: This is a multicentre, double-blind, randomised controlled study to determine the optimal dose and duration of treatment for the correction of vitamin D insufficiency or deficiency in patients with CKD5d; to investigate whether vitamin D supplementation delays the increase in PTH levels in this group of patients; and to investigate the effects on changes in CKD-MBD-related markers, cardiovascular complications, cognitive function in this group of patients. 2. Study procedure: Based on the inclusion and exclusion of the patients, the study was conducted in accordance with the following criteria
2. Study procedure: Eligible subjects were screened according to inclusion and exclusion criteria and randomly divided into three groups: high-dose vitamin D group, low-dose vitamin D group and control group. Baseline data were collected before the intervention and each group was given different doses of regular vitamin D2 softgels or placebo and followed up. 25(OH)D, PTH, blood Ca, and blood P levels were measured every month; bone metabolism markers, FGF23, and blood counts, liver function, kidney function, lipids, and blood glucose were measured every 3 months; the prevalence of vascular calcification, the incidence of cardiovascular events, and changes in cognitive function scale scores were assessed 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with chronic kidney disease stage 5d who have been on haemodialysis for 3 months or more
3. 5 ng/mL < 25(OH)D < 30 ng/mL (liquid phase tandem mass spectrometry).
4. 130 pg/ml < PTH < 600 pg/ml (electrochemiluminescence method).
5. serum phosphorus < 1.78 mmol/L.
6. Good compliance with the treatment requirements formulated for the study.
7. informed consent from the subject.

Exclusion Criteria:

1. Patients who are prepped for or have undergone renal transplantation or parathyroidectomy.
2. taking vitamin D, active vitamin D or analogues and other drugs that may affect 25(OH)D levels within 3 months prior to enrolment
3. Treatment affecting PTH results (e.g. cenacaser, etc.) within 3 months prior to enrolment
4. Serum calcium > 2.55 mmol/L
5. Patients who are pregnant or likely to become pregnant, breastfeeding or planning to become pregnant during the study period
6. known prior or concomitant serious illness or medical condition such as malignancy, human immunodeficiency virus, severe gastrointestinal or liver disease, intestinal malabsorptive disease, hepatitis or cardiovascular events that may worsen or shorten life expectancy and/or interfere with participation in the study
7. History of neurological/psychiatric disease, including psychosis or dementia, or any other reason that is unlikely to result in adherence to treatment or follow-up plans.
8. Known or suspected allergy to any component of the study drug.
9. Ongoing participation in other clinical studies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Differences in changes in PTH levels from baseline to 6 months of intervention | baseline，at 6 months intervention

SECONDARY OUTCOMES:
Differences in changes in PTH levels from baseline to intervention at 1months、2months、3months、4months、5months | baseline，at 1，2，3，4，5 months intervention
Proportion of 25(OH)D >30ng/ml at 3 months of intervention | at 3 months intervention
Trends in changes in 25(OH)D levels from baseline to intervention at 1months、2months、3months、4months、5months、6months | baseline，at 1，2，3，4，5，6 months intervention
Incidence of cardiovascular events after 6 months of intervention | baseline，at 6 months intervention
Change in prevalence of vascular calcification at 6 months of intervention | baseline，at 6 months intervention
  We used cardiac ultrasound and lateral abdominal views to look for vascular calcification
Change in Montreal Cognitive Assessment Scale scores at 6 months of intervention | baseline，at 6 months intervention
  A total score of 30 on this scale, with a score of ≥26 indicating normal; a score of <26 indicates the presence of cognitive impairment: 18-26 for mild cognitive impairment, 10-17 for moderate cognitive impairment and <10 for severe cognitive impairment
Trends in blood calcium levels at 1 month, 2 months, 3 months, 4 months, 5 months and 6 months of intervention | baseline，at 1，2，3，4，5，6 months intervention
Trends in blood phosphorus levels at 1 month, 2 months, 3 months, 4 months, 5 months and 6 months of intervention | baseline，at 1，2，3，4，5，6 months intervention
Trends in FGF23 levels at 3 and 6 months of intervention | baseline，at 3，6 months intervention
Trends in Osteocalcin(OC) levels at 3 and 6 months of intervention | baseline，at 3，6 months intervention
Trends in Precollagen type I amino-terminal peptide(PINP) levels at 3 and 6 months of intervention | baseline，at 3，6 months intervention
Trends in β specific collagen degradation products(β-CTX) levels at 3 and 6 months of intervention | baseline，at 3，6 months intervention
Trends in ALP levels at 3 and 6 months of intervention | baseline，at 3，6 months intervention
Incidence of fractures at 6 months of intervention | baseline，at 6 months intervention
  Ask if the patient had a fracture during the intervention, the site of the fracture and the type of fracture
Incidence of falls at 6 months of intervention | baseline，at 6 months intervention
  Ask if the patient has fallen during the intervention, the number of falls and the reasons for them

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The data including baseline characteristics of study population, blood biochemical index and main outcome measures may be made available.
Supporting Information: Study Protocol, SAP